CLINICAL TRIAL: NCT01664104
Title: CRP and BMI Study: Evaluation in Real Life of Clinical Remission Rate and Correlation Between CRP and BMI in Patients Treated With Tocilizumab
Brief Title: A Study to Evaluate Tocilizumab Treatment in a Real-Life Setting
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28336
Record Dates: First submitted 2012-08-07; First posted 2012-08-14 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- RA Participants: Participants with moderate or severe RA who are under tocilizumab treatment in routine clinical practice (in accordance with the local label) will be observed for 6 months from the start of treatment.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be administered in routine clinical practice in accordance with local label. Study protocol does not specify/enforce any treatment regimen.

SUMMARY:
This observational, multi-center study will evaluate the treatment regimen, treatment responses and safety of tocilizumab therapy in a routine clinical practice in participants with moderate to severe rheumatoid arthritis (RA). Data will be collected for 6 months with a maximum study duration of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe RA according to revised American College of Rheumatology criteria
* Participants have started tocilizumab treatment according to routine clinical practice within 3 months prior to site opening and still in treatment, as well as participants who began treatment at enrollment

Exclusion Criteria:

* Participants who have started tocilizumab treatment more than 3 months prior to site opening
* Participants who have previously received tocilizumab in a clinical trial setting or for compassionate use
* Participants who have been enrolled in an ongoing clinical trial and/or have received treatment with any investigational drug within 4 weeks prior to study start
* Participants with a history of autoimmune disease or joint inflammatory disease other than RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate to severe RA who are being treated or begin treatment with tocilizumab according to routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- Italy (22):
  - Coppito, Abruzzo
  - Barletta, Apulia
  - Casarano (LE), Apulia
  - Foggia, Apulia
  - Reggio Calabria, Calabria
  - Benevento, Campania
  - Telese Terme, Campania
  - Bologna, Emilia-Romagna
  - Rome, Lazio
  - Bergamo, Lombardy
  - Castel Goffredo, Lombardy
  - Gavardo, Lombardy
  - Milan, Lombardy
  - Monza, Lombardy
  - Pavia, Lombardy
  - Novara, Piedmont
  - Catania, Sicily
  - Palermo, Sicily
  - Florence, Tuscany
  - Pisa, Tuscany
  - Cona (Ferrara), Veneto
  - Verona, Veneto

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 151 participants were enrolled in the study; of which,136 participants met the eligibility criteria. The results are reported only for those participants who met the eligibility criteria.
Groups:
- Rheumatoid Arthritis (RA) Participants: Participants with moderate or severe RA who were under tocilizumab (TCZ) treatment in routine clinical practice (in accordance with the local label) were observed for 6 months from the start of treatment.
Period: Overall Study
Arm/Group | Rheumatoid Arthritis (RA) Participants
Started | 136
Completed | 120
Not Completed | 16
Not completed — Adverse Event | 6
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 4
Not completed — Other | 1
Not completed — Unknown: Reason Unrelated to TCZ | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants evaluable for primary objective: All enrolled participants except participants who withdrew from study for reasons not related to TCZ and had not interrupted TCZ treatment at withdrawal; lost to follow-up participants in treatment with TCZ at withdrawal; or premature termination occurring until 5 months from start of TCZ.
Groups:
- RA Participants: Participants with moderate or severe RA who were under TCZ treatment in routine clinical practice (in accordance with the local label) were observed for 6 months from the start of treatment.
Arm/Group | RA Participants
Number analyzed (Participants) | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on TCZ Treatment at Month 6
Description: Percentage of participants on TCZ treatment at Month 6 was calculated as: [(participants on TCZ treatment at Month 6) divided by (participants evaluable for primary objective)] multiplied by 100. Confidence interval was computed based on the Clopper-Pearson method.
Time Frame: Month 6
Population: All enrolled participants evaluable for primary objective.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 133
percentage of participants | 86.5 [79.46 to 91.78]

2. Secondary Outcome: Percentage of Participants by TCZ Dose at Month 6
Description: TCZ dose at Month 6 was calculated over the total number of participants evaluable for the primary objective and who did not interrupt TCZ. Percentage of participants on TCZ dose at Month 6 was calculated as the [(participants with specified TCZ dose at 6 months) divided by (participants who did not interrupt TCZ at Month 6)] multiplied by 100.
Time Frame: Month 6
Population: All enrolled participants evaluable for primary objective and who did not interrupt TCZ at Month 6.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 115
percentage of participants
  8 milligrams per kilogram (mg/kg) | 93.91
  4 mg/kg | 1.74
  6.35 mg/kg | 0.87
  7.1 mg/kg | 0.87
  7.6 mg/kg | 0.87
  6.4 mg/kg | 0.87
  Not available | 0.87

3. Secondary Outcome: Percentage of Participants Starting TCZ After Inadequate Response (IR) to a Biologic Treatment or After Intolerance or IR to Disease-Modifying Anti-Rheumatic Drugs (DMARDs)
Description: Participants with at least 1 treatment with biologic agent not equal missing and which is not ongoing or with a stop date lower or equal to first TCZ administration had IR to biologic treatment. Participants with at least 1 treatment with DMARDs with a stop date lower or equal to first TCZ administration had IR to DMARDs. Participants with a biologic and DMARDs interruption or with a biologic interruption and ongoing treatment with DMARDs were classified in "IR to biologic group". Participants with DMARDs interruption or ongoing DMARDs and adding TCZ without a biologic interruption were classified in the "DMARDs intolerance and/or IR" group.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 133
percentage of participants
  IR to biologic treatment | 62.4
  Intolerance or IR to DMARDs | 37.6

4. Secondary Outcome: Time Elapsed From Diagnosis of RA
Description: Time elapsed from diagnosis of RA in years was calculated as the (difference between the date of enrollment visit and the date of first diagnosis of RA) divided by 365.25.
Time Frame: Baseline (assessed retrospectively)
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Median (Full Range); unit: years
Arm/Group | RA Participants
Number analyzed (Participants) | 131
years | 6.5 [0.3 to 49.5]

5. Secondary Outcome: Patient Assessment of Pain Using Visual Analog Scale (VAS) at Baseline
Description: Participants measured the pain intensity due to RA on a 100 millimeter (mm) VAS, where the responses were on a continuous range from 0 mm = no pain to 100 mm = unbearable pain.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants
Number analyzed (Participants) | 125
mm | 61.3 (28.2)

6. Secondary Outcome: Patient Global Assessment of Disease Activity (PGH) Using VAS at Baseline
Description: The PGH was measured using a 100 mm VAS, where the responses were on a continuous range from 0 mm = managing very well to 100 mm = managing very poorly.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants
Number analyzed (Participants) | 117
mm | 61.0 (28.5)

7. Secondary Outcome: Physician Global Assessment of Disease Activity (PhGH) Using VAS at Baseline
Description: The PhGH was measured on a 100 mm VAS, where 0 mm = no arthritis activity to 100 mm = extremely active arthritis.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants
Number analyzed (Participants) | 114
mm | 53.4 (24.6)

8. Secondary Outcome: Participant Assessment of Morning Stiffness Using VAS at Baseline
Description: The participant assessment of morning stiffness was measured using a ruler on a 100 mm VAS, where the responses were on a continuous range from 0 mm = no stiffness and 100 mm = maximum stiffness.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants
Number analyzed (Participants) | 50
mm | 47.0 (32.6)

9. Secondary Outcome: Participant Assessment of Fatigue Using VAS at Baseline
Description: Participants measured the level of fatigue due to RA using a 100 mm VAS, where the responses were on a continuous range from 0 mm = no fatigue to 100 mm = extreme fatigue.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants
Number analyzed (Participants) | 91
mm | 57.1 (29.0)

10. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Baseline
Description: The HAQ-DI is a questionnaire that measures functional status (disability) and health-related quality of life (QoL). It measures the participant's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common activities over past week. Each question was evaluated according to the degree of severity on a 4-point scale ranging from 0 = without any difficulty to 3 = unable to do. Total score for HAQ-DI is the average of all questions and ranges from 0 to 3, where higher scores represent higher disease activity.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 111
units on a scale | 1.4 (0.6)

11. Secondary Outcome: Tender Joint Count (TJC) at Baseline
Description: TJC was determined by examining 28 joints and identifying the joints that were painful under pressure or to passive motion. Tenderness was recorded on the joint assessment form at baseline; no tenderness = 0 and tenderness = 1.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | RA Participants
Number analyzed (Participants) | 130
tender joints | 11.5 (7.5)

12. Secondary Outcome: Swollen Joint Count (SJC) at Baseline
Description: SJC was determined by examining 28 joints and identifying when swelling was present. Swelling was recorded on the joint assessment form at baseline; no swelling = 0 and swelling = 1.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | RA Participants
Number analyzed (Participants) | 130
swollen joints | 6.7 (5.5)

13. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) at Baseline
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeter per hour (mm/hour). A decrease in the level indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | RA Participants
Number analyzed (Participants) | 131
mm/hour | 33.0 (25.1)

14. Secondary Outcome: C-Reactive Protein (CRP) at Baseline
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | RA Participants
Number analyzed (Participants) | 126
milligrams per deciliter (mg/dL) | 2.7 (7.9)

15. Secondary Outcome: Percentage of Participants With Presence of Extra-Articular Systemic Features of RA at Baseline
Description: Extra-articular systemic features referred to anemia, fatigue as well as a wide range of co-morbidities such as osteoporosis and other iatrogenic complications. Percentage of participants with any of the extra-articular systemic feature are reported.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- RA Participants: Participants with moderate or severe RA were prescribed with tocilizumab, in accordance with routine clinic practice, and following the local label were observed for 6 months with maximum study duration of 18 months.
Arm/Group | RA Participants
Number analyzed (Participants) | 128
percentage of participants | 7.0

16. Secondary Outcome: Percentage of Participants With Evidence of Structural Joint Damage at Baseline
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 114
percentage of participants | 71.9

17. Secondary Outcome: Percentage of Participants With Previous RA-Related Surgical Procedures at Baseline
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 124
percentage of participants | 12.9

18. Secondary Outcome: Percentage of Participants With Positive Rheumatoid Factor (RF) at Baseline
Description: RF is the auto antibody directed against immunoglobulin G and its concentration is observed in human serum or plasma. RF value higher than 20 units per milliliter is considered positive.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 116
percentage of participants | 59.5

19. Secondary Outcome: Percentage of Participants With Anti-Citrullinated Cyclic Peptide at Baseline
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 103
percentage of participants | 58.3

20. Secondary Outcome: Percentage of Participants by Duration of Morning Stiffness at Baseline
Description: Duration of morning stiffness was defined as the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was able to resume normal activities without stiffness. The participant reported the duration of morning stiffness in the case report form by ticking 1 of the following categories: no morning stiffness, less than (<) 30 minutes, 30 - 60 minutes, 60 - 120 minutes, 120 - 240 minutes, greater than (>) 240 minutes, and the whole day. 'Not estimable' represented that the participants were not able to quantify it.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 133
percentage of participants
  No morning stiffness | 6.8
  < 30 minutes | 15.0
  Between 30 - 60 minutes | 30.1
  Between 60 - 120 minutes | 25.6
  Between 120 - 240 minutes | 4.5
  > 240 minutes | 3.8
  The whole day | 2.3
  Not estimable | 12.0

21. Secondary Outcome: Number of Participants With TCZ Dose Change According to the Reason for Change
Description: Number of participants with TCZ dose change (increase or decrease with respect to starting dose) was reported by reason for change.
Time Frame: Baseline up to Month 6
Population: All enrolled participants evaluable for the primary objective and had TCZ dose modification.
Measure: Number; unit: participants
Arm/Group | RA Participants
Number analyzed (Participants) | 6
participants
  Adverse event | 3
  Physician decision | 1
  Weight variation | 1
  Other | 1

22. Secondary Outcome: Percentage of Participants by Number of TCZ Dose Modifications Per Participant
Description: The number of TCZ dose modifications per participant was calculated as the number of times that the participant changed the prescribed dose with respect to the dose planned at enrollment/previous administration. If the participant did not change the prescribed dose, the values were set at missing.
Time Frame: Baseline up to Month 6
Population: All enrolled participants evaluable for primary objective.
Measure: Number; unit: percentage of participants
Groups:
- RA Participants: Participants with moderate or severe RA who were prescribed with tocilizumab, in accordance with routine clinic practice, and following the local label were observed for 6 months with maximum study duration of 18 months.
Arm/Group | RA Participants
Number analyzed (Participants) | 133
percentage of participants
  0 dose modification | 95.49
  1 dose modification | 1.50
  2 dose modifications | 3.01

23. Secondary Outcome: Time in Days Elapsed Between TCZ Infusions
Description: The time elapsed in days between TCZ infusions was calculated as the difference between the date of TCZ infusion and the date of the previous administration.
Time Frame: Baseline up to Month 6 (assessed retrospectively and prospectively at each administration [approximately 1 month apart] up to administration 8
Population: All enrolled participants evaluable for primary objective. Here, Number of participants analyzed = participants evaluable for the outcome measure and number analyzed = participants with available data for specified category.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | RA Participants
Number analyzed (Participants) | 130
days
  Infusion 1 and Infusion 2 | 31 [28 to 35]
  Infusion 2 and Infusion 3: number analyzed (Participants) | 124
  Infusion 2 and Infusion 3 | 31.5 [28.5 to 34]
  Infusion 3 and Infusion 4: number analyzed (Participants) | 121
  Infusion 3 and Infusion 4 | 31 [28 to 35]
  Infusion 4 and Infusion 5: number analyzed (Participants) | 115
  Infusion 4 and Infusion 5 | 30 [28 to 35]
  Infusion 5 and Infusion 6: number analyzed (Participants) | 107
  Infusion 5 and Infusion 6 | 31 [28 to 35]
  Infusion 6 and Infusion 7: number analyzed (Participants) | 79
  Infusion 6 and Infusion 7 | 29 [28 to 33]
  Infusion 7 and Infusion 8: number analyzed (Participants) | 15
  Infusion 7 and Infusion 8 | 28 [28 to 31]

24. Secondary Outcome: Percentage of Participants With TCZ Infusion Interruption
Description: The percentage of participants with at least one infusion interruption was reported as "Yes". Participants with unknown infusion interruption were set to "No".
Time Frame: Baseline up to Month 6
Population: All enrolled participants evaluable for primary objective.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 133
percentage of participants
  Yes | 3.01
  No | 96.99

25. Secondary Outcome: Percentage of Participants Who Discontinued TCZ by Reason for Discontinuation
Time Frame: Baseline up to Month 6
Population: All enrolled participants evaluable for primary objective who discontinued TCZ.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 18
percentage of participants
  Adverse event | 50.0
  Lack of or insufficient efficacy | 33.33
  Unspecified | 16.67

26. Secondary Outcome: Percentage of Participants With TCZ Reintroduction
Description: The percentage of participants with at least one TCZ reintroduction was reported as "Yes". Participants with unknown TCZ reintroduction were set to "No".
Time Frame: Baseline up to Month 6
Population: All enrolled participants evaluable for primary objective.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 133
percentage of participants
  Yes | 1.5
  No | 98.5

27. Secondary Outcome: Percentage of Participants by Reason for Choice of TCZ Monotherapy at Baseline
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 40
percentage of participants
  Lack of DMARD efficacy | 12.5
  DMARD intolerability | 85
  Both lack of efficacy and intolerability to DMARDs | 2.5

28. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28 Joint Count (DAS28) Score at Month 3 and Month 6
Description: DAS28 score is a measurement of RA activity on a 0 to 10 scale, with higher scores representing higher disease activity, and calculated as DAS28 = 0.56 x √TJC28 + 0.28 x √SJC28 + 0.36 x natural logarithm (ln) (CRP + 1) + 0.014 x PGH + 0.96, where TJC28 = tender joint count on 28 units, SJC28 = swollen joint count on 28 units, CRP = serum concentration of c-reactive protein (after converting units to mg/dL), PGH = patient global assessment of disease activity, which was measured on a 100 mm VAS, where 0 mm = managing very well and 100 mm = managing very poorly (√ = square root). A score of < 2.6 represents clinical remission, a score of greater than or equal to (≥) 2.6 and less than or equal to (≤) 3.2 represents low disease activity, a score of > 3.2 and ≤ 5.1 represents moderate disease activity and a score of > 5.1 represents high (or severe) disease activity. Change from baseline = DAS28 at Month X - DAS28 at baseline. Here X = 3 and 6 for Change at Months 3 and 6, respectively.
Time Frame: Baseline, Month 3, and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 37
units on a scale
  Baseline | 5.16 (1.06)
  Change at Month 3 | 1.99 (1.04)
  Change at Month 6 | 2.15 (1.26)
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon test — P-value was calculated between baseline versus change at Month 3
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon test — P-value was calculated between baseline versus change at Month 6

29. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) Score at Month 3 and Month 6
Description: SDAI is a combined index for measuring disease activity in RA and calculated as SDAI = TJC28 + SJC28 + PGH (in cm) + PhGH (in cm) + CRP (in mg/dL), where TJC28 = tender joint count on 28 units, SJC28 = swollen joint count on 28 units, PGH = patient's global assessment of disease activity, assessed on a 100 mm VAS, where 0 = managing very well and 100 = managing very poorly, PhGH = physician global assessment of disease activity, assessed on a 100 mm VAS, where 0 mm = no arthritis activity and 100 mm = extremely active arthritis, CRP = serum concentration of C-reactive protein. SDAI total score ranged from 0-86. Higher scores represent greater disease activity. SDAI scores of ≤ 3.3 represents clinical remission, ≤ 11.0 represents low disease activity , ≤ 26.0 represents moderate disease activity, and > 26.0 represents high (or severe) disease activity. Change from baseline = SDAI score at Month X - SDAI score at baseline. Here X = 3 and 6 for Change at Months 3 and 6, respectively.
Time Frame: Baseline, Month 3, and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 61
units on a scale
  Baseline | 35.12 (20.50)
  Change at Month 3 | 19.37 (17.08)
  Change at Month 6 | 20.35 (22.00)
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon test — P-value was calculated between baseline versus change at Month 3
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon test; P-value was calculated between baseline versus change at Month 6

30. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score at Month 3 and Month 6
Description: The CDAI is a combined index for measuring disease activity in RA and calculated as CDAI = TJC28 + SJC28 + PGH (in cm) + PhGH (in cm), where TJC28 = tender joint count on 28 units, SJC28 = swollen joint count on 28 units, PGH = patient's global assessment of disease activity, assessed on a 100 mm VAS, where 0 = managing very well and 100 = managing very poorly, and PhGH = physician global assessment of disease activity, assessed on a 100 mm VAS, where 0 mm = no arthritis activity and 100 mm = extremely active arthritis. CDAI total score ranged from 0-76. Higher scores indicate greater disease activity. CDAI score of ≤ 2.8 represents clinical remission, score of ≤ 10.0 represents low disease activity, score of ≤ 22.0 represents moderate disease activity, and score of > 22.0 represents high (or severe) disease activity. Change from baseline = CDAI score at Month X - CDAI score at baseline. Here X = 3 and 6 for Change at Months 3 and 6, respectively.
Time Frame: Baseline, Month 3, and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 80
units on a scale
  Baseline | 30.48 (13.62)
  Change at Month 3 | 15.06 (13.56)
  Change at Month 6 | 15.96 (15.73)
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon test; P-value was calculated between baseline versus change at Month 3
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon test; P-value was calculated between baseline versus change at Month 6

31. Secondary Outcome: Percentage of Participants by DAS28 Class at the Start of TCZ Treatment and After Month 3 and Month 6
Description: DAS28 score is a measurement of RA activity on a 0 to 10 scale and calculated as DAS28 = 0.56 x √TJC28 + 0.28 x √SJC28 + 0.36 x ln(CRP + 1) + 0.014 x PGH + 0.96, where TJC28 = tender joint count on 28 units, SJC28 = swollen joint count on 28 units, CRP = serum concentration of c-reactive protein (after converting units to mg/dL), PGH = patient's global assessment of disease activity, which was measured on a 100 mm VAS, where 0 mm = managing very well and 100 mm = managing very poorly. Higher scores represent greater disease activity. A score of < 2.6 represents clinical remission, a score of ≥ 2.6 and ≤ 3.2 represents low disease activity, a score of >3.2 and ≤ 5.1 represents moderate disease activity, and a score of > 5.1 represents high (or severe) disease activity.
Time Frame: Baseline, Month 3, and Month 6
Population: All enrolled participants evaluable for primary objective. Here, Number of participants analyzed= participants evaluable for this outcome and number analyzed = participants with available data for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 92
percentage of participants
  Baseline: DAS28 < 2.6: number analyzed (Participants) | 57
  Baseline: DAS28 < 2.6 | 3.5
  Baseline: DAS28 ≥ 2.6 to ≤ 3.2: number analyzed (Participants) | 57
  Baseline: DAS28 ≥ 2.6 to ≤ 3.2 | 1.8
  Baseline: DAS28 > 3.2 to ≤ 5.1: number analyzed (Participants) | 57
  Baseline: DAS28 > 3.2 to ≤ 5.1 | 43.9
  Baseline: DAS28 > 5.1: number analyzed (Participants) | 57
  Baseline: DAS28 > 5.1 | 50.9
  Month 3: DAS28 < 2.6 | 30.4
  Month 3: DAS28 ≥ 2.6 to ≤ 3.2 | 14.1
  Month 3: DAS28 >3.2 to ≤ 5.1 | 50.0
  Month 3: DAS28 > 5.1 | 5.4
  Month 6: DAS28 < 2.6: number analyzed (Participants) | 86
  Month 6: DAS28 < 2.6 | 33.7
  Month 6: DAS28 ≥ 2.6 to ≤ 3.2: number analyzed (Participants) | 86
  Month 6: DAS28 ≥ 2.6 to ≤ 3.2 | 15.1
  Month 6: DAS28 >3.2 to ≤ 5.1: number analyzed (Participants) | 86
  Month 6: DAS28 >3.2 to ≤ 5.1 | 43.0
  Month 6: DAS28 > 5.1: number analyzed (Participants) | 86
  Month 6: DAS28 > 5.1 | 8.1

32. Secondary Outcome: Percentage of Participants by SDAI Class at the Start of TCZ Treatment and After Month 3 and Month 6
Description: SDAI is a combined index for measuring disease activity in RA and calculated as SDAI = TJC28 + SJC28 + PGH (in cm) + PhGH (in cm) + CRP (in mg/dL), where TJC28 = tender joint count on 28 units, SJC28 = swollen joint count on 28 units, PGH = patient's global assessment of disease activity, assessed on a 100 mm VAS, where 0 mm = managing very well and 100 mm = managing very poorly, PhGH = physician global assessment of disease activity, assessed on a 100 mm VAS, where 0 = no arthritis activity and 100 = extremely active arthritis, CRP = serum concentration of C-reactive protein. SDAI total score ranged from 0-86. Higher scores represent greater disease activity. SDAI scores of ≤ 3.3 represents clinical remission, ≤ 11.0 represents low disease activity, ≤ 26.0 represents moderate disease activity, and > 26.0 represents high (or severe) disease activity.
Time Frame: Baseline, Month 3, and Month 6
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 93
percentage of participants
  Baseline: SDAI ≤ 3.3 | 2.2
  Baseline: SDAI ≤ 11.0 | 7.5
  Baseline: SDAI ≤ 26.0 | 36.6
  Baseline: SDAI > 26.0 | 63.4
  Month 3: SDAI ≤ 3.3: number analyzed (Participants) | 83
  Month 3: SDAI ≤ 3.3 | 7.2
  Month 3: SDAI ≤ 11.0: number analyzed (Participants) | 83
  Month 3: SDAI ≤ 11.0 | 34.9
  Month 3: SDAI ≤ 26.0: number analyzed (Participants) | 83
  Month 3: SDAI ≤ 26.0 | 80.7
  Month 3: SDAI > 26.0: number analyzed (Participants) | 83
  Month 3: SDAI > 26.0 | 19.3
  Month 6: SDAI ≤ 3.3: number analyzed (Participants) | 80
  Month 6: SDAI ≤ 3.3 | 13.8
  Month 6: SDAI ≤ 11.0: number analyzed (Participants) | 80
  Month 6: SDAI ≤ 11.0 | 47.5
  Month 6: SDAI ≤ 26.0: number analyzed (Participants) | 80
  Month 6: SDAI ≤ 26.0 | 82.5
  Month 6: SDAI > 26.0: number analyzed (Participants) | 80
  Month 6: SDAI > 26.0 | 17.5

33. Secondary Outcome: Percentage of Participants by CDAI Class at the Start of TCZ Treatment and After Month 3 and Month 6
Description: CDAI is a combined index for measuring disease activity in RA and calculated as CDAI = TJC28 + SJC28 + PGH (in cm) + PhGH (in cm), where TJC28 = tender joint count on 28 units, SJC28 = swollen joint count on 28 units, PGH = patient's global assessment of disease activity, assessed on a 100 mm VAS, where 0 mm = managing very well and 100 mm = managing very poorly, and PhGH = physician global assessment of disease activity, assessed on a 100 mm VAS, where 0 mm = no arthritis activity and 100 mm = extremely active arthritis. CDAI total score ranged from 0-76. Higher scores indicate greater disease activity. CDAI score of ≤ 2.8 represents clinical remission, score of ≤ 10.0 represents low disease activity, score of ≤ 22.0 represents moderate disease activity, and score of > 22.0 represents high (or severe) disease activity.
Time Frame: Baseline, Month 3, and Month 6
Population: All enrolled participants evaluable for primary objective. Here, Number of participants analyzed= participants evaluable for the outcome measure and number analyzed = participants with available data for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 97
percentage of participants
  Baseline: CDAI ≤ 2.8 | 2.1
  Baseline: CDAI ≤ 10.0 | 8.2
  Baseline: CDAI ≤ 22.0 | 24.7
  Baseline: CDAI > 22.0 | 75.3
  Month 3: CDAI ≤ 2.8: number analyzed (Participants) | 94
  Month 3: CDAI ≤ 2.8 | 7.4
  Month 3: CDAI ≤ 10.0: number analyzed (Participants) | 94
  Month 3: CDAI ≤ 10.0 | 36.2
  Month 3: CDAI ≤ 22.0: number analyzed (Participants) | 94
  Month 3: CDAI ≤ 22.0 | 77.7
  Month 3: CDAI > 22.0: number analyzed (Participants) | 94
  Month 3: CDAI > 22.0 | 22.3
  Month 6: CDAI ≤ 2.8: number analyzed (Participants) | 94
  Month 6: CDAI ≤ 2.8 | 10.6
  Month 6: CDAI ≤ 10.0: number analyzed (Participants) | 94
  Month 6: CDAI ≤ 10.0 | 42.6
  Month 6: CDAI ≤ 22.0: number analyzed (Participants) | 94
  Month 6: CDAI ≤ 22.0 | 78.7
  Month 6: CDAI > 22.0: number analyzed (Participants) | 94
  Month 6: CDAI > 22.0 | 21.3

34. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20%, 50%, 70%, or 90% (ACR20/50/70/90) Response After Month 3 and Month 6 From the Start of TCZ Treatment
Description: ACR20, 50, 70 or 90 response = an improvement of ≥20%, ≥50%, ≥70% or ≥90% respectively, as compared to baseline in TJC28 and SJC28, and 20/50/70/90%, improvement in at least 3 of 5 following measures: Patient's Assessment of Pain over previous 24 hours, PGH, PhGH, HAQ, and acute phase reactant (either CRP or ESR). TJC and SJC, based on 28-joint assessments. Number of tender joints and swollen joints were recorded on joint assessment form at baseline; no tenderness = 0 and tenderness = 28, no swelling = 0 and swelling = 28, respectively. HAQ measures functional status (disability) and health-related QoL with 20 questions, summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common activities over past week, 0= without difficulty to 3= unable to do. Patient's assessment of pain assessed using VAS; 0 mm = no pain, 100 mm = unbearable pain; PGH and PhGH, assessed using VAS; 0 mm = no disease activity, 100 mm = maximum disease activity.
Time Frame: Month 3 and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 120
percentage of participants
  Month 3: ACR 20 achieved | 45
  Month 3: ACR 20 not achieved | 38.3
  Month 3: ACR 20 at least 1 missing data | 16.7
  Month 3: ACR 50 achieved | 23.3
  Month 3: ACR 50 not achieved | 62.5
  Month 3: ACR 50 at least 1 missing data | 14.2
  Month 3: ACR 70 achieved | 9.2
  Month 3: ACR 70 not achieved | 79.2
  Month 3: ACR 70 at least 1 missing data | 11.7
  Month 3: ACR 90 achieved | 1.7
  Month 3: ACR 90 not achieved | 90.0
  Month 3: ACR 90 at least 1 missing data | 8.3
  Month 6: ACR 20 achieved | 51.7
  Month 6: ACR 20 not achieved | 35.8
  Month 6: ACR 20 at least 1 missing data | 12.5
  Month 6: ACR 50 achieved | 27.5
  Month 6: ACR 50 not achieved | 57.5
  Month 6: ACR 50 at least 1 missing data | 15.0
  Month 6: ACR 70 achieved | 12.5
  Month 6: ACR 70 not achieved | 73.3
  Month 6: ACR 70 at least 1 missing data | 14.2
  Month 6: ACR 90 achieved | 2.5
  Month 6: ACR 90 not achieved | 89.2
  Month 6: ACR 90 at least 1 missing data | 8.3

35. Secondary Outcome: Change From Baseline to Month 6 in TJC
Description: TJC was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at baseline and at Month 6. No tenderness = 0 and tenderness = 1.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | RA Participants
Number analyzed (Participants) | 114
tender joints | 6.0 (7.9)

36. Secondary Outcome: Change From Baseline to Month 6 in SJC
Description: SJC was determined by examination of 28 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at baseline and at Month 6. No swelling = 0 and swelling = 1.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | RA Participants
Number analyzed (Participants) | 114
swollen joints | 4.2 (6.1)

37. Secondary Outcome: Change From Baseline to Month 6 in PGH
Description: The PGH was measured using a 100 mm VAS, where the responses were on a continuous range from 0 mm = managing very well and 100 mm = managing very poorly.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for the primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants
Number analyzed (Participants) | 96
mm | 21.4 (26.1)

38. Secondary Outcome: Change From Baseline to Month 6 in PhGH
Description: The PhGH was evaluated using a 100 mm VAS where 0 mm = no arthritis activity and 100 mm = extremely active arthritis. Higher scores indicated increased level of disease.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for the primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants
Number analyzed (Participants) | 93
mm | 23.9 (26.2)

39. Secondary Outcome: Change From Baseline to Month 6 in Patient's Assessment of Pain
Description: Participants measured the pain intensity due to RA using a 100 mm VAS, where the responses were on a continuous range from 0 mm = no pain to 100 mm = unbearable pain.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants
Number analyzed (Participants) | 107
mm | 22.5 (26.4)

40. Secondary Outcome: Change From Baseline to Month 6 in HAQ-DI Score
Description: The HAQ-DI is a questionnaire that measures functional status (disability) and health-related QoL. It measures the participant's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common activities over past week. Each question was evaluated according to the degree of severity on a 4-point scale ranging from 0 = without any difficulty to 3 = unable to do.Total score for HAQ-DI is the average of all the questions, which ranges from 0 to 3, where higher scores represent higher disease activity.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for the primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 89
units on a scale | 0.4 (0.6)

41. Secondary Outcome: Change From Baseline to Month 6 in Participant Assessment of Fatigue
Description: as for outcome 9
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for the primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants
Number analyzed (Participants) | 68
mm | 17.9 (23.1)

42. Secondary Outcome: Change From Baseline to Month 6 in Participant Assessment of Morning Stiffness
Description: as for outcome 8
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants
Number analyzed (Participants) | 35
mm | 18.8 (31.6)

43. Secondary Outcome: Percentage of Participants With Clinically Meaningful Improvement in HAQ-DI
Description: The HAQ-DI is a questionnaire that measures functional status (disability) and health-related QoL. It measures the participant's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common activities over past week. Each question was evaluated according to the degree of severity on a 4-point scale ranging from 0 = without any difficulty to 3 = unable to do. Total score for HAQ-DI is the average of all the questions, which ranges from 0 to 3, where higher scores represent higher disease activity. HAQ-DI clinically meaningful improvement is defined as decrease in HAQ total score from baseline of greater or equal to 0.22 points.
Time Frame: Month 3 and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 120
percentage of participants
  Month 3 | 36.7
  Month 6 | 45.8

44. Secondary Outcome: Percentage of Participants Achieving Good/Moderate/No European League Against Rheumatism (EULAR) Response at Month 3 and Month 6
Description: Clinical response was assessed according to EULAR criteria that classified the participant according to individual changes in DAS28 score as good, moderate, or no response. DAS28 score is a measurement of RA activity on 0 to 10 scale and calculated as DAS28= 0.56 x √TJC28 + 0.28 x √SJC28 + 0.36 x ln(CRP + 1) + 0.014 x PGH + 0.96, where TJC28= tender joint count on 28 units, SJC28= swollen joint count on 28 units, CRP= serum concentration of C-reactive protein (after converting units to mg/dL), PGH= patient's global assessment of disease activity measured on a 100 mm VAS, where 0 mm= managing very well and 100 mm= managing very poorly. Good responders experienced change (chg) from baseline (BL) of >1.2 with DAS28 score ≤ 3.2, moderate responders experienced chg from BL >1.2 with DAS28 score > 3.2 to ≤ 5.1 or a chg from BL > 0.6 to ≤ 1.2 with DAS28 score of ≤ 5.1. No responders experienced chg from BL < 0.6 regardless initial DAS28 score or > 0.6 to ≤ 1.2 with DAS28 score of > 5.1.
Time Frame: Month 3 and Month 6
Population: as for outcome 33
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 46
percentage of participants
  Month 3: Good response | 41.3
  Month 3: Moderate response | 47.8
  Month 3: No response | 10.9
  Month 6: Good response: number analyzed (Participants) | 44
  Month 6: Good response | 45.5
  Month 6: Moderate response: number analyzed (Participants) | 44
  Month 6: Moderate response | 40.9
  Month 6: No response: number analyzed (Participants) | 44
  Month 6: No response | 13.6

45. Secondary Outcome: Time to DMARD Dose Reduction
Description: DMARDs that met the criteria for "concomitant medications" were selected. The time to DMARD dose reduction was calculated as the difference between date of dose reduction and the date of first TCZ infusion. For participants presenting more than 1 DMARD dose reduction, only the first dose reduction was considered.
Time Frame: Baseline up to Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | RA Participants
Number analyzed (Participants) | 9
months | 3.2 [1.0 to 4.6]

46. Secondary Outcome: Time to DMARD Dose Withdrawal
Description: DMARDs that met the criteria for "concomitant medications" were selected. The time to DMARD withdrawal was calculated as the difference between date of withdrawal and the date of first TCZ infusion.
Time Frame: Baseline up to Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | RA Participants
Number analyzed (Participants) | 11
months | 4.1 [2.9 to 5.2]

47. Secondary Outcome: Percentage of Participants by Reason for DMARD Withdrawal During the Study
Description: DMARDs that met the criteria for "concomitant medications" were selected. All treatments with DMARDs interrupted after the first TCZ infusion were selected.
Time Frame: Baseline up to Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 11
percentage of participants
  Lack of efficacy | 18.18
  Subjective intolerance | 9.09
  Objective intolerance | 36.36
  Unspecified | 36.36

48. Secondary Outcome: Time to Steroid Dose Reduction
Description: Steroids that met the criteria for "concomitant medications" were selected. The time to steroid dose reduction was calculated as the difference between date of dose reduction and the date of first TCZ infusion. For participants presenting more than one steroid dose reduction, only the first dose reduction was considered.
Time Frame: Baseline up to Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | RA Participants
Number analyzed (Participants) | 18
months | 2.3 [1.7 to 4.6]

49. Secondary Outcome: Time to Steroid Dose Withdrawal
Description: Steroids that met the criteria for "concomitant medications" were selected. The time to steroid dose withdrawal was calculated as the difference between date of withdrawal and the date of first TCZ infusion.
Time Frame: Baseline up to Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | RA Participants
Number analyzed (Participants) | 7
months | 1.8 [1.1 to 3.1]

50. Secondary Outcome: Change From Baseline in CRP at Month 3 and Month 6
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. Change from baseline = CRP level at Month X - CRP level at baseline. Here X = 3 and 6 for Change at Months 3 and 6, respectively.
Time Frame: Baseline, Month 3, and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | RA Participants
Number analyzed (Participants) | 89
mg/dL
  Change at Month 3 | 2.28 (8.61)
  Change at Month 6 | 1.98 (8.87)
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon test — P-value was calculated between baseline versus change at Month 3
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon test — P-value was calculated between baseline versus change at Month 6

51. Secondary Outcome: Change From Baseline in ESR at Month 3 and Month 6
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hr. A decrease in the level indicates reduction in inflammation and therefore improvement. Change from baseline = ESR level at Month X - ESR level at baseline. Here X = 3 and 6 for Change at Months 3 and 6, respectively.
Time Frame: Baseline, Month 3, and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | RA Participants
Number analyzed (Participants) | 100
mm/hr
  Change at Month 3 | 23.15 (21.72)
  Change at Month 6 | 21.42 (23.21)
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon test — P-value was calculated between baseline versus change at Month 3
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon test — P-value was calculated between baseline versus change at Month 6

52. Secondary Outcome: CRP at the Start of TCZ Treatment by Remission Status Using DAS28-CRP, SDAI, and CDAI at Month 6
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. DAS28 is calculated as follows: DAS28 = 0.56 x √TJC28 + 0.28 x √SJC28 + 0.36 x ln(CRP + 1) + 0.014 x PGH + 0.96, A score of < 2.6 represents clinical remission. SDAI is a combined index for measuring disease activity in RA and calculated as SDAI = TJC28 + SJC28 + PGH (in cm) + PhGH (in cm) + CRP (in mg/dL). A SDAI score of ≤ 3.3 represents clinical remission. CDAI is a combined index for measuring disease activity in RA and calculated as CDAI = TJC28 + SJC28 + PGH (in cm) + PhGH (in cm). A CDAI score of ≤ 2.8 represents clinical remission.
Time Frame: Baseline
Population: All enrolled participants evaluable for primary objective. Here, Number of participants analyzed = participants evaluable for this outcome measure and number analyzed = participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | RA Participants
Number analyzed (Participants) | 89
mg/dL
  With DAS28-CRP clinical remission: number analyzed (Participants) | 27
  With DAS28-CRP clinical remission | 2.2 (6.2)
  Without DAS28-CRP clinical remission: number analyzed (Participants) | 54
  Without DAS28-CRP clinical remission | 3.1 (10.5)
  With SDAI clinical remission: number analyzed (Participants) | 9
  With SDAI clinical remission | 4.6 (10.6)
  Without SDAI clinical remission: number analyzed (Participants) | 66
  Without SDAI clinical remission | 2.8 (9.5)
  With CDAI clinical remission: number analyzed (Participants) | 10
  With CDAI clinical remission | 4.2 (10.0)
  Without CDAI clinical remission: number analyzed (Participants) | 79
  Without CDAI clinical remission | 2.7 (8.8)
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p = 0.6904, t-test; P-value signifies CRP at the start of TCZ treatment by remission status using DAS28-CRP (remission versus no remission)
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p = 0.6032, t-test; P-value signifies the CRP at the start of TCZ treatment by remission status using SDAI (remission versus no remission)
Statistical Analysis 3: Comparison: RA Participants; Test type: Superiority or Other; p = 0.6146, t-test; P-value signifies the CRP at the start of TCZ treatment by remission status using CDAI (remission versus no remission)

53. Secondary Outcome: Body Mass Index (BMI) at the Start of TCZ Treatment by Remission Status Using DAS-28 CRP, SDAI, and CDAI at Month 6
Description: DAS28 scale ranges from 0 to 10, and calculated as DAS28 = 0.56 x √TJC28 + 0.28 x √SJC28 + 0.36 x ln(CRP + 1) + 0.014 x PGH + 0.96, where TJC28 and SJC28 = tender joint and swollen joint count on 28 units, PGH = patient's global assessment of disease activity, assessed on a 100 mm VAS, where 0 mm = managing very well and 100 mm = managing very poorly, CRP = serum concentration of C-reactive protein. A score of < 2.6 represents clinical remission. SDAI is a combined index for measuring disease activity in RA and calculated as SDAI = TJC28 + SJC28 + PGH (in cm) + PhGH (in cm) + CRP (in mg/dL), where PhGH = physician global assessment of disease activity, assessed on a 100 mm VAS, where 0 mm = no arthritis activity and 100mm = extremely active arthritis. A SDAI score of ≤ 3.3 represents clinical remission. CDAI is a combined index for measuring disease activity in RA and calculated as CDAI = TJC28 + SJC28 + PGH (in cm) + PhGH (in cm). A CDAI score of ≤ 2.8 represents clinical remission.
Time Frame: Baseline
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: kilogram per meter square (Kg/m^2)
Arm/Group | RA Participants
Number analyzed (Participants) | 91
kilogram per meter square (Kg/m^2)
  With DAS-28 CRP clinical remission: number analyzed (Participants) | 26
  With DAS-28 CRP clinical remission | 23.3 (3.2)
  Without DAS-28 CRP clinical remission: number analyzed (Participants) | 57
  Without DAS-28 CRP clinical remission | 26.7 (5.0)
  With SDAI clinical remission: number analyzed (Participants) | 10
  With SDAI clinical remission | 23.7 (3.2)
  Without SDAI clinical remission: number analyzed (Participants) | 68
  Without SDAI clinical remission | 26.0 (5.0)
  With CDAI clinical remission: number analyzed (Participants) | 10
  With CDAI clinical remission | 23.8 (3.3)
  Without CDAI clinical remission: number analyzed (Participants) | 81
  Without CDAI clinical remission | 26.6 (5.8)
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p = 0.0018, t-test; P-value signifies the BMI at the start of TCZ treatment by remission status using DAS28-CRP (remission versus no remission)
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p = 0.1617, t-test; P-value signifies the BMI at the start of TCZ treatment by remission status using SDAI (remission versus no remission)
Statistical Analysis 3: Comparison: RA Participants; Test type: Superiority or Other; p = 0.1296, t-test; P-value signifies the BMI at the start of TCZ treatment by remission status using CDAI (remission versus no remission)

54. Secondary Outcome: Percentage of Participants With and Without Morning Stiffness
Description: Morning stiffness was defined by the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was able to resume normal activities without stiffness. The participant assessed morning stiffness based on the following criteria:
  1. Presence of participant's joints stiff when woke up that day, measured as yes (stiffness present) or no (stiffness not present);
  2. Duration of morning stiffness, measured by ticking 1 of the six categories: < 30 minutes, 30 - 60 minutes, 60 - 120 minutes, 120 - 240 minutes, > 240 minutes, and the whole day;
  3. Severity of morning stiffness measured using a ruler on a 100 mm VAS where the responses were on a continuous range from 0 mm = no stiffness to 100 mm = maximum stiffness.
  'Not estimable' represented that the participants were not able to quantify it. 'Not done' represented that the assessment was not performed.
Time Frame: Month 3 and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 120
percentage of participants
  Month 3 (with morning stiffness) | 70.0
  Month 3 (without morning stiffness) | 15.8
  Month 3 (morning stiffness not estimable) | 10.8
  Month 3 (morning stiffness not done) | 3.3
  Month 6 (with morning stiffness) | 65.0
  Month 6 (without morning stiffness) | 25.8
  Month 6 (morning stiffness not estimable) | 9.2

55. Secondary Outcome: Percentage of Participants by Duration of Morning Stiffness
Description: Duration of morning stiffness was defined as the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was able to resume normal activities without stiffness. The participant reported the duration of morning stiffness in the case report form by ticking 1 of the following categories: no morning stiffness, < 30 minutes, 30 - 60 minutes, 60 - 120 minutes, 120 - 240 minutes, > 240 minutes, and the whole day. 'Not estimable' represented that the participants were not able to quantify it. 'Not done' represented that the assessment was not performed.
Time Frame: Month 3 and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 120
percentage of participants
  Month 3 (no morning stiffness) | 15.8
  Month 6 (no morning stiffness) | 25.8
  Month 3 (< 30 minutes) | 40.8
  Month 6 (< 30 minutes) | 35.0
  Month 3 (between 30 - 60 minutes ) | 20.0
  Month 6 (between 30 - 60 minutes) | 21.7
  Month 3 (Between 60 - 240 minutes) | 7.5
  Month 6 (Between 60 - 240 minutes) | 7.5
  Month 3 (> 240 minutes) | 0.8
  Month 6 (> 240 minutes) | 0
  Month 3 (whole day) | 0
  Month 6 (whole day) | 0.8
  Month 3 (not estimable) | 11.7
  Month 6 (not estimable) | 9.2
  Month 3 (not done) | 3.3

56. Secondary Outcome: CRP at the Start of TCZ Treatment by Morning Stiffness at Month 6
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. The participant reported the duration of morning stiffness in the case report form by ticking the categories: ≤ 30 minutes and > 30 minutes.
Time Frame: Baseline
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | RA Participants
Number analyzed (Participants) | 40
mg/dL
  Morning stiffness (≤ 30 minutes) | 3.3 (12.0)
  Morning stiffness (> 30 minutes): number analyzed (Participants) | 39
  Morning stiffness (> 30 minutes) | 2.1 (2.9)
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p = 0.5332, t-test; P-value signifies the CRP at the start of TCZ treatment using the morning stiffness ( ≤ 30 minutes versus > 30 minutes)

57. Secondary Outcome: BMI at the Start of TCZ Treatment by Morning Stiffness at Month 6
Description: Morning stiffness was defined as the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was able to resume normal activities without stiffness. The participant reported the duration of morning stiffness in the case report form by ticking the categories: ≤ 30 minutes and > 30 minutes.
Time Frame: Baseline
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | RA Participants
Number analyzed (Participants) | 39
Kg/m^2
  Morning stiffness (≤ 30 minutes) | 26.1 (4.0)
  Morning stiffness (> 30 minutes): number analyzed (Participants) | 37
  Morning stiffness (> 30 minutes) | 26.6 (5.9)
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p = 0.6159, t-test; P-value signifies the BMI at the start of TCZ treatment using the morning stiffness ( ≤ 30 minutes versus > 30 minutes)

58. Secondary Outcome: Correlation Coefficient Between CRP (mg/dL) at the Start of TCZ Treatment and HAQ-DI (0-3) at Month 6
Description: The test for CRP is laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in level of CRP indicates reduction in inflammation and therefore improvement. HAQ-DI is a questionnaire that measures functional status (disability) and health-related QoL. It measures the participant's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common activities over past week. Each question was evaluated according to the degree of severity on a 4-point scale ranging from 0 = without any difficulty to 3 = unable to do. Total score is average of all questions, which ranges from 0 to 3, where higher scores represent higher disease activity. The Pearson and Spearman correlation coefficients can range in value from -1 to +1.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: correlation coefficient
Arm/Group | RA Participants
Number analyzed (Participants) | 89
correlation coefficient
  Pearson correlation | 0.12663
  Spearman correlation | 0.02678
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p = 0.2370, Pearson correlation; P-value was calculated from Pearson correlation coefficient between CRP at the start of TCZ treatment versus HAQ-DI (0-3) at Month 6
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p = 0.8033, Spearman Correlation; P-value was calculated from Spearman correlation coefficient between CRP at the start of TCZ treatment versus HAQ-D1 (0-3) at Month 6

59. Secondary Outcome: Correlation Coefficient Between Change From Baseline in CRP (mg/dL) and HAQ-DI (0-3) at Month 6
Description: CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in level of CRP indicates reduction in inflammation and therefore improvement. HAQ-DI is a questionnaire that measures functional status (disability) and health-related QoL. It measures the participant's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common activities over past week. Each question was evaluated according to the degree of severity on a 4-point scale ranging from 0= without any difficulty to 3= unable to do. Total score is the average of all questions, which ranges from 0 to 3, where higher scores represent higher disease activity. The Pearson and Spearman correlation coefficients can range in value from -1 to +1.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: correlation coefficient
Arm/Group | RA Participants
Number analyzed (Participants) | 72
correlation coefficient
  Pearson correlation | 0.25513
  Spearman correlation | 0.21125
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p = 0.0306, Pearson correlation; P-value was calculated from Pearson correlation coefficient for change from baseline in CRP versus change from baseline in HAQ-DI (0-3) at Month 6
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p = 0.0749, Spearman Correlation; P-value was calculated from Spearman correlation coefficient for change from baseline in CRP versus change from baseline in HAQ-DI (0-3) at Month 6

60. Secondary Outcome: Correlation Coefficient Between CRP (mg/dL) at the Start of TCZ Treatment and VAS Fatigue at Month 6
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. Participants measured the level of fatigue due to RA using a 100 mm VAS, where the responses were on a continuous range from 0 mm = no fatigue to 100 mm = extreme fatigue. The Pearson and Spearman correlation coefficients can range in value from -1 to +1.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: correlation coefficient
Arm/Group | RA Participants
Number analyzed (Participants) | 75
correlation coefficient
  Pearson correlation | 0.08180
  Spearman correlation | -0.11521
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p = 0.4854, Pearson correlation; P-value was calculated from Pearson correlation coefficient between CRP at the start of TCZ treatment versus VAS fatigue at Month 6
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p = 0.3250, S; P-value was calculated from Spearman correlation coefficient between CRP at the start of TCZ treatment versus VAS fatigue at Month 6

61. Secondary Outcome: Correlation Coefficient Between Change From Baseline in CRP (mg/dL) at the Start of TCZ Treatment and Change From Baseline in VAS Fatigue at Month 6
Description: as for outcome 60
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: correlation coefficient
Arm/Group | RA Participants
Number analyzed (Participants) | 59
correlation coefficient
  Pearson correlation | 0.41350
  Spearman correlation | 0.40842
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p = 0.0011, Pearson correlation; P-value was calculated from Pearson correlation coefficient between change from baseline in CRP versus change from baseline in VAS fatigue at Month 6
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p = 0.0013, Spearman Correlation; P-value calculated from Spearman correlation coefficient between change from baseline in CRP versus change from baseline in VAS fatigue at Month 6

62. Secondary Outcome: Correlation Coefficient Between BMI at the Start of TCZ Treatment and HAQ-DI (0-3) at Month 6
Description: The HAQ-DI is a questionnaire that measures functional status (disability) and health-related QoL. It measures the participant's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene,reach, grip and common activities over past week. Each question was evaluated according to the degree of severity on a 4-point scale ranging from 0 = without any difficulty to 3 = unable to do. Total score is the average of all questions, which ranges from 0 to 3, where higher scores represent higher disease activity. The Pearson and Spearman correlation coefficients can range in value from -1 to +1.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: correlation coefficient
Arm/Group | RA Participants
Number analyzed (Participants) | 48
correlation coefficient
  Pearson correlation | 0.08505
  Spearman correlation | 0.12488
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p = 0.5655, Pearson correlation; P-value was calculated from Pearson correlation coefficient between BMI at the start of TCZ treatment versus HAQ-DI (0-3) at Month 6
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p = 0.3977, Spearman Correlation; P-value was calculated from Spearman correlation coefficient between BMI at the start of TCZ treatment versus HAQ-DI (0-3) at Month 6

63. Secondary Outcome: Correlation Coefficient Between Change From Baseline in CRP (mg/dL) and Change From Baseline in Morning Stiffness According to VAS at Month 6
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. Morning stiffness was defined as the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was able to resume normal activities without stiffness. The participant reported the duration of morning stiffness in the case report form by ticking 1 of the following categories: no morning stiffness, < 30 minutes, 30 - 60 minutes, 60 - 120 minutes, 120 - 240 minutes, > 240 minutes, and the whole day. The Pearson and Spearman correlation coefficients can range in value from -1 to +1.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: correlation coefficient
Arm/Group | RA Participants
Number analyzed (Participants) | 35
correlation coefficient
  Pearson correlation | 0.41875
  Spearman correlation | 0.40754
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p = 0.0123, Pearson correlation; P-value obtained from Pearson correlation coefficient between change from baseline in CRP versus change from baseline in morning stiffness at Month 6
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p = 0.0151, Spearman Correlation; P-value obtained from Spearman correlation coefficient between change from baseline in CRP versus change from baseline in morning stiffness at Month 6

64. Secondary Outcome: Correlation Coefficient Between BMI at the Start of TCZ Treatment and VAS Fatigue at Month 6
Description: Participants measured the level of fatigue due to RA using a 100 mm VAS, where the responses were on a continuous range from 0 mm = no fatigue to 100 mm = extreme fatigue. The Pearson and Spearman correlation coefficients can range in value from -1 to +1.
Time Frame: Baseline and Month 6
Population: All enrolled participants evaluable for primary objective with available data for this outcome measure.
Measure: Number; unit: correlation coefficient
Arm/Group | RA Participants
Number analyzed (Participants) | 42
correlation coefficient
  Pearson correlation | 0.00181
  Spearman correlation | -0.07250
Statistical Analysis 1: Comparison: RA Participants; Test type: Superiority or Other; p = 0.9909, Pearson correlation; P-value was calculated from Pearson correlation coefficient between BMI at the start of TCZ treatment versus VAS fatigue at Month 6
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p = 0.6482, Spearman Correlation; P-value was calculated from Spearman correlation coefficient between BMI at the start of TCZ treatment versus VAS fatigue at Month 6

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from enrollment up to 6 months (final visit).
Description: Safety Analysis Set: Participants evaluable at enrollment.
Arm/Group | RA Participants
Serious Adverse Events (participants affected / at risk) | 2/136
Other Adverse Events (participants affected / at risk) | 8/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RA Participants (N=136)
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RA Participants (N=136)
Cough (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.